CLINICAL TRIAL: NCT02820207
Title: Vascular Surgery Department of Beijing Tsinghua Chang Gung Hospital
Brief Title: Identification of Carotid Plague Vulnerability by Contrast Enhanced Ultrasound: Correlation With Plague Histopathology
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Keqiang Zhao, Attending Doctor, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: （2016）003
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2020-07

CONDITIONS: Carotid Artery Plaque; Ultrasonic Diagnosis
Keywords: Carotid Artery Plaque; Contrast Enhanced Ultrasound; Plague Histopathology
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vulnerable plague: The patients suffering from carotid artery stenosis were identified as the vulnerable plague group by Contrast Enhanced Ultrasound whose plagues were found intraplaque neovascularization

SUMMARY:
OBJECTIVE/BACKGROUND: Intraplaque neovascularization is one of the most important risk factors for unstable carotid plaque. This study was designed to evaluate whether carotid intraplaque neovascularization (IPN) can be accurately assessed by contrast enhanced ultrasound (CEUS).

METHODS: Preoperative CEUS analysis of 50 carotid artery stenosis patients would be compared to histopathology performed on their plaques excised by carotid endarterectomy (CEA) with CD34 and MMP9 staining.

DETAILED DESCRIPTION:
1. To enroll 50 cases of patients suffering from carotid artery stenosis continuously, the investigators perform contrast enhanced ultrasound on patients for identifying the vulnerable plagues and taking high resolution MR inspection to analysis those plagues at the same time.
2. All patients undergo carotid endarterectomy. The vulnerable ingredients of carotid plaques such as intraplaque neovascularization and bleeding are identified by pathological examination and immunohistochemical staining.
3. To evaluate the accuracy of CEUS for identifying carotid vulnerable plague compared with high resolution MR.
4. The investigators divide patients into the stable group and the vulnerable group based on the results of CEUS inspection. To analysis the incidence of postoperative complications such as stroke and mortality within 30 days and to compare the differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients with ischemic symptom whose carotid stenosis were more than 50%
* The patients without ischemic symptom whose carotid stenosis were more than 70%

Exclusion Criteria:

* Confirmed with severe intracranial vascular lesions
* Suffering from the large area cerebral infarction or critical stroke sequela
* Restenosis after CEA or CAS
* Suffering from severe coronary heart disease, respiratory failure,the hypertension difficult to controled
* Patients with malignant tumor or expected life < 2 years

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients suffering from carotid artery stenosis
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
the incidence of ischemia shock | within 30 days after operations
  The incidence of ischemic stroke was defined as the number of cases of postoperative cerebral infarction divided by the total number of cases

SECONDARY OUTCOMES:
the incidence of restenosis | 6 months after operations
  the loss of lumen of carotid beyond 70% is defined as restenosis
the incidence of all-cause mortality | within 30 days after operations
  All-cause mortality includes all causes of death, such as MI, heart failure, stroke, bleeding et al.

CONTACTS AND LOCATIONS:
Overall Officials: sifan Yang, M.D., Study Director — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No